CLINICAL TRIAL: NCT05280431
Title: Evaluation of the Use of Exoskeleton Systems for Upper Limb Rehabilitation in Neurological Patients
Brief Title: Evaluation of Exoskeleton for Upper Limb Rehabilitation in Neurological Patients
Acronym: PCP_EXOs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Casa di Cura Privata del Policlinico SpA (Other)
Collaborators: Politecnico di Milano (Other); Fundación Tecnalia Research & Innovation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PCP_EXOs_
Record Dates: First submitted 2022-02-10; First posted 2022-03-15 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-02

CONDITIONS: Stroke; Neurologic Disorder
MeSH Terms: conditions — Stroke; Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (AGREE) (Experimental): 15 sessions, 3 sessions per week. Each session consists of 45 minutes of training with the AGREE exoskeleton. The training session is customized to the patient's needs and can be adapted to his/her improvement during the intervention.
  Interventions: Device: AGREE exoskeleton
- Experimental Group (FEXO) (Experimental): 15 sessions, 3 sessions per week. Each session consists of 45 minutes of training with the FEXO exoskeleton. The training session is customized to the patient's needs and can be adapted to his/her improvement during the intervention.
  Interventions: Device: FEXO exoskeleton
- Control Group (Conventional therapy) (Other): 15 sessions, 3 sessions per week. Each session consists of 45 minutes and consists of different training modalities typically used in the rehabilitation of the arm after stroke.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: AGREE exoskeleton — Upper limb exoskeleton with four actuated degrees of freedom (shoulder horizontal adduction/abduction, shoulder flexion/extension, humeral rotation, elbow flexion/extension), and one passive degree of freedom (wrist pronation/supination), implementing different rehabilitative strategies.
  The intervention consists of the execution of different exercises with the affected arm supported by the AGREE device. The subject is actively involved in the exercises and the system provides different kinds of assistance that can be tailored according to the patient's status.
  The following exercises can be performed:
  * anterior reaching (in a plane or in the space)
  * lateral elevation of the arm
  * hand to mouth movements with or without an object in the hand
  * moving objects (on a plane or in the space)
  * exergames.
  A subset of exercises is defined based on the patient's capability.
  Arms: Experimental Group (AGREE)
Device: FEXO exoskeleton — After patient's preparation (tDCS and FES) the FEXO assessment is conducted. The subject performs FEXO assessment games. This stage is also used to calibrate the reach and grasp movement intention EEG patterns. The movement is recorded using internal kinematic sensors; therefore, these measures can be extracted for both reaching and lifting movements. Trunk forward bending is measured to avoid compensatory movements when doing reaching assessment. The clinician then reviews the plan for today's session: game selection, number of repetitions and assistance levels. The patient gets ready to play the games and the clinician starts the first activity of the active stage of FEXO therapy. The patient plays the game and sees his own results. The clinician monitors patient activity, assistance levels, effort and signs of discomfort. The patient plays the next game and sees his own results, and the clinician checks the patient's progress with the results overview.
  Arms: Experimental Group (FEXO)
Other: Conventional therapy — It consists of a combination of different treatment modalities among the following, based on the patient's specific needs:
  * Upper limb passive motion
  * Occupational therapy exercises
  * Constraint-induced movement therapy
  * Upper limb active movement (reaching, grasping, elevation, spatial orientation)
  * Repetitive task training
  Arms: Control Group (Conventional therapy)

SUMMARY:
Acquired cerebrovascular trauma is the third most common cause of disability worldwide, resulting in long-term disability, limitation of activities of daily living, and reduced social participation. It is estimated that, within three months of the acute event, a high percentage of patients do not recover full function. 93% of these disabilities concern the upper limb.

To induce optimal functional reorganization after the acute cerebrovascular events or neurodegenerative diseases affecting the central nervous system, robotic assistance allows intensive exercises with specific therapeutic purposes. Indeed, they enable an intensive, repetitive, and customizable therapeutic program that is in line with the principles underlying motor learning.

Clinical investigation is needed to assess the efficacy of the proposed new technologies (AGREE and FEXO exoskeleton) and to guide subsequent developmental steps. Therefore, an exploratory clinical study is proposed to evaluate usability, tolerability, and safety, as well as to assess the effectiveness of the new technologies.

The primary objective of this study is to examine the safety and tolerability of the new active exoskeletons for upper extremity rehabilitation and validate them in a controlled environment. Furthermore, efficacy will be examined as the secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 85 years;
* motor deficit of the upper limb induced by neurological diseases (e.g., stroke, multiple sclerosis);
* time since the acute event of at least one month;
* Trunk Control Test score ≥ 48.

Exclusion Criteria:

* global aphasia;
* presence of cognitive impairment;
* severe unilateral spatial neglect;
* Box and Block test < 1;
* Ashworth scale score ≥ 4;
* total or severe impairment of visual acuity;
* instability of clinical parameters or presence of severe comorbidities;
* inadequate anthropometric measurements;
* presence of any serious condition that may affect participation in the study (e.g., oncological, hepatic/renal, immune, metabolic/endocrine, psychiatric, respiratory or infectious disorders);
* inability to comply with the protocol or to give informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | up to 5 weeks
  SUS is used to measure how easy or difficult the proposed system is to use

SECONDARY OUTCOMES:
Technology Assessment Methods (TAM) | up to 5 weeks
  TAM is an information systems theory that models how users come to accept and use a technology
Virtual Reality Questionnaire (VR) | up to 5 weeks
  VR is used to measure how easy or difficult the virtual reality interface is to use
Fugl-Meyer Assessment Scale (FMA-UE) | up to 5 weeks
  FMA-UE assesses sensorimotor status including items assessing upper extremity motion, balance, sensation and range of movement
Action Research Arm Test (ARAT) | up to 5 weeks
  ARAT is used to assess upper extremity performance (coordination, dexterity and functioning)
Modified Ashworth Scale (MAS) | up to 5 weeks
  MAS is used to muscle quantified spasticity
Motricity Index (MI) | up to 5 weeks
  MI is used to grade motor activity in muscles of the upper limb
Visual Analogue Scale (VAS) | up to 5 weeks
  VAS is a psychometric response scales used to measure subjective pain
Box and Block Test (BBT) | up to 5 weeks
  BBT measures unilateral gross manual dexterity. The BBT administration consists of asking the subject to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds
Nine Hole Peg Test (9HPT) | up to 5 weeks
  9HPT is used to measure finger dexterity in patients. The 9HPT administration consist of asking the subject to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible
Number of Peaks (#Peaks) of the speed profile | up to 5 weeks
  If a point-to-point reaching movement has a low number of peaks, it means that few acceleration and deceleration periods are present
Smoothness described by the Teulings's index (TI) | up to 5 weeks
  TI s the rate of change of the acceleration in a movement; a lower value of TI indicates a smoother movement
The absolute hand path error (e) | up to 5 weeks
  e is the area between the actual movement path and the straight line; this was considered an index of learning and a reduction of e indicates a better adaptation to the required task.
Event-Related Desynchronization and Synchronization (ERD/ERS) of the μ and β rhythms | up to 5 weeks
  Motor processing can result in changes of the ongoing EEG in form of an event-related desynchronization (ERD) or event-related synchronization (ERS). Spatial mapping of ERD/ERS can be used to study the dynamics of cortical activation patterns

CONTACTS AND LOCATIONS:
Locations (1):
- Casa di Cura del Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No